CLINICAL TRIAL: NCT01902693
Title: Prospective Observational Study of HIV Positive Individuals on Suppressive HAART With Malignancy Undergoing Chemotherapy
Brief Title: Prospective HIV Chemotherapy Cohort Study
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRO2009; CHERUB 003-301 (Other Grant/Funding Number: Imperial Biomedical Research Centre award)
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: HIV; Cancer
Keywords: HIV; Chemotherapy; Cohort; Cancer; HAART; Malignancy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV & chemotherapy: Participants will be aged ≥ 18 years, aware of their HIV status and the diagnosis of malignancy, have a plasma viral load of < 50 HIV-1 RNA copies/ml (on suppressive HAART) at enrolment and be designated to receive cytotoxic chemotherapy including one or more of the following agents: R-CHOP, ABVD, Liposomal doxorubicin (Caelyx) or liposomal daunorubicin (Daunoxome) or Paclitaxel.
  There is no intervention for this study. Blood samples will be taken and if available from routine care surplus cerebrospinal fluid.
  Interventions: Other: No intervention for this study

INTERVENTIONS:
Other: No intervention for this study — No intervention

SUMMARY:
Human Immunodeficiency Virus (HIV) infection is very successfully treated with a type of therapy called Highly Active AntiRetroviral Therapy (HAART). Although HAART has made a great improvement to the health and lives of all people living with HIV, HAART cannot be stopped because it is not able to 'cure' or eliminate the HIV virus from all cells in the body - the remaining viruses are referred to as 'latent' or sleeping virus. As soon as the HAART treatment is stopped the virus comes back (wakes up). It is for this reason that stopping HAART treatment is not recommended. However, it may be that other drugs if given with HAART could have a stronger effect on the latent virus. There is some evidence from laboratory research that suggests that some of the drugs we use to treat certain types of cancer may have an effect on the latent virus. The purpose of this research study is to use new laboratory research technology to measure the amount of 'latent' virus in people who are treated with HAART who then need to use chemotherapy treatments for cancer. We will look at whether the levels of HIV virus are reduced in patients having chemotherapy by looking at the virus levels before, during and after chemotherapy treatment. We do not know very much about how HIV persists in the body despite therapy and unless new approaches are developed, removal of the HIV virus from all cells in the body will not be possible.

DETAILED DESCRIPTION:
STUDY DESIGN This study will be performed at one investigational site in the UK. This is a single centre, prospective observational cohort study of HIV positive individuals on suppressive HAART with malignancy undergoing chemotherapy.

ELIGIBILITY Individuals receiving HAART and diagnosed with either lymphoma or Kaposi's sarcoma receiving combination chemotherapy agents, which include the vinca alkaloids and taxanes, will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and able to give written informed consent
* Be aware of their HIV status and the diagnosis of malignancy
* Have a plasma viral load of < 50 HIV-1 RNA copies/ml (on suppressive HAART) at enrolment
* Be designated to receive cytotoxic chemotherapy including one or more of the following agents: R-CHOP, ABVD, Liposomal doxorubicin (Caelyx) or liposomal daunorubicin (Daunoxome) or Paclitaxel

Exclusion Criteria:

* Patients not receiving HAART
* A detectable (>50 HIV-1 RNA copies/ml) HIV plasma viral load at screening
* Opportunistic infections
* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited only from Chelsea and Westminster joint HIV oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proviral DNA | 12 weeks postcompletion of chemotherapy
  Comparison of proviral DNA quantification between baseline and at 12 weeks postcompletion of chemotherapy

SECONDARY OUTCOMES:
Proviral DNA | Baseline, prior to mid cycle of chemotherapy, prior to the final cycle of chemotherapy, 4 weeks post chemotherapy and 12 weeks post chemotherapy
  Quantification of proviral DNA (intracellular DNA/MRNA)
Viral RNA | Baseline, prior to mid cycle of chemotherapy, prior to the final cycle of chemotherapy, 4 weeks post chemotherapy and 12 weeks post chemotherapy
  Quantification of HIV-1 viral RNA transcripts
Ultra-low viral load | Baseline, prior to mid cycle of chemotherapy, prior to the final cycle of chemotherapy, 4 weeks post chemotherapy and 12 weeks post chemotherapy
  Quantification of HIV-1 ultra-low viral load (UL-VL)
Immune activation levels | Baseline, prior to mid cycle of chemotherapy, prior to the final cycle of chemotherapy, 4 weeks post chemotherapy and 12 weeks post chemotherapy
  Quantification of immune activation levels
Histone deacetylase inhibition | Baseline, prior to mid cycle of chemotherapy, prior to the final cycle of chemotherapy, 4 weeks post chemotherapy and 12 weeks post chemotherapy
  Degree of histone deacetylase inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fidler, Principal Investigator — Imperial College London
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom